CLINICAL TRIAL: NCT07277231
Title: A Phase 3, Open-Label, Randomized Study of Sonrotoclax (BGB-11417) Plus Zanubrutinib (BGB-3111) Compared With Venetoclax Plus Acalabrutinib in Patients With Previously Untreated Chronic Lymphocytic Leukemia
Brief Title: A Study to Investigate Sonrotoclax (BGB-11417) Plus Zanubrutinib (BGB-3111) Compared With Venetoclax Plus Acalabrutinib in Adults With Previously Untreated Chronic Lymphocytic Leukemia
Status: Not yet recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: BeOne Medicines (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: BGB-11417-304; 2025-524366-21-00 (EU CTIS Number)
Record Dates: First submitted 2025-12-02; First posted 2025-12-11 (Actual); Last update posted 2025-12-11 (Actual); Status verified 2025-12

CONDITIONS: Chronic Lymphocytic Leukemia
Keywords: B-cell Lymphoma-2 Inhibitor; Bruton Tyrosine Kinase Inhibitor
MeSH Terms: conditions — Leukemia, Lymphocytic, Chronic, B-Cell | interventions — zanubrutinib; acalabrutinib; venetoclax

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Arm A: Sonrotoclax plus Zanubrutinib (Experimental): Participants will receive sonrotoclax and zanubrutinib for a fixed duration followed by observation.
  Interventions: Drug: Sonrotoclax; Drug: Zanubrutinib
- Arm B: Venetoclax plus Acalabrutinib (Active Comparator): Participants will receive venetoclax and acalabrutinib for a fixed duration followed by observation.
  Interventions: Drug: Acalabrutinib; Drug: Venetoclax

INTERVENTIONS:
Drug: Sonrotoclax — Administered orally.
  Other Names: BGB-11417
  Arms: Arm A: Sonrotoclax plus Zanubrutinib
Drug: Zanubrutinib — Administered orally.
  Other Names: BGB-3111; Brukinsa
  Arms: Arm A: Sonrotoclax plus Zanubrutinib
Drug: Acalabrutinib — Administered orally.
  Other Names: Calquence
  Arms: Arm B: Venetoclax plus Acalabrutinib
Drug: Venetoclax — Administered orally.
  Other Names: Venclexta; Venclyxto
  Arms: Arm B: Venetoclax plus Acalabrutinib

SUMMARY:
The purpose of this study is to investigate the efficacy and safety of fixed-duration sonrotoclax (also known as BGB-11417) plus zanubrutinib (also known as BGB-3111) (SZ) compared with fixed-duration of venetoclax plus acalabrutinib (AV) in participants with previously untreated chronic lymphocytic leukemia (CLL).

ELIGIBILITY:
Inclusion Criteria:

* Treatment-naïve (TN) adults with confirmed diagnosis of CLL which requires treatment
* Eastern Cooperative Oncology Group (ECOG) score 0, 1, or 2
* Measurable disease by Computer Tomography/Magnetic Resonance Imaging
* Adequate bone marrow and organ function

Exclusion Criteria:

* Previous systemic treatment for CLL
* Known prolymphocytic leukemia or history of, or currently suspected, Richter's transformation
* Known central nervous system involvement
* History of confirmed progressive multifocal leukoencephalopathy (PML)
* Uncontrolled hypertension or clinically significant cardiovascular disease

Note: Other protocol defined Inclusion/Exclusion criteria may apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 500 (Estimated)
Dates: Start 2026-01-31 (Estimated); Primary Completion 2031-02 (Estimated); Study Completion 2031-11 (Estimated)

PRIMARY OUTCOMES:
Progression-Free Survival (PFS) as Determined by Independent Review Committee (IRC) | Up to approximately 70 months
  PFS is defined as the time from the date of randomization to the date of disease progression as determined by IRC or death due to any cause, whichever occurs first.
Rate of Undetectable Minimal Residual Disease at < 10^-4 sensitivity (uMRD4) | Up to approximately 16 months
  Rate of uMRD4 is defined as the percentage of participants that achieved uMRD4 measured in both peripheral blood (PB) and bone marrow aspirate (BMA) at the post-treatment follow-up visit (PTFU1) based on next generation sequencing (NGS).

SECONDARY OUTCOMES:
PFS in High-Risk Participants | Up to approximately 70 months
  PFS is defined as the time from the date of randomization to the date of disease progression as determined by IRC or death due to any cause, whichever occurs first.
Overall Survival (OS) | Up to approximately 70 months
  OS is defined as the time from the date of randomization to the date of death due to any cause.
Overall Response Rate (ORR) as Determined by IRC | Up to approximately 70 months
  ORR is defined as the percentage of participants with a complete response (CR), complete response with incomplete hematopoietic recovery (CRi), nodal partial response (nPR), or partial response (PR), before disease progression, death, or the start of new anti-CLL treatment (whichever is earlier), as assessed by IRC.
Rate of Undetectable Minimal Residual Disease at < 10^-5 sensitivity (uMRD5) | Up to approximately 16 months
  Rate of uMRD5 is defined as the percentage of participants who achieved uMRD5 measured in both PB and BMA at the PTFU1 Visit based on NGS, before disease progression, death, or the start of new anti-CLL treatment (whichever is earlier).
Number of Participants with Adverse Events | Up to approximately 70 months
  Number of participants with treatment-emergent adverse events (TEAEs), adverse events of clinical interest, and serious adverse events (SAEs), including laboratory values, vital signs, and physical examination findings.
PFS Determined by Investigator Assessment | Up to approximately 70 months
  PFS is defined as the time from the date of randomization to the date of disease progression as determined by investigator or death due to any cause, whichever occurs first.
Complete Response Rate (CRR) by IRC and Investigator Assessment | Up to approximately 70 months
  CRR is defined as the percentage of participants with a CR or CRi before disease progression, death, or the start of new anti-CLL treatment (whichever is earlier).
ORR Determined by Investigator Assessment | Up to approximately 70 months
  ORR is defined as the percentage of participants with a complete response or partial response, before disease progression, death, or the start of new anti-CLL treatment (whichever is earlier), as assessed by investigator.
Duration of Response (DOR) | Up to approximately 70 months
  Duration of response (determined by both IRC and investigator assessment) is defined as the time from the first qualifying response (CR, CRi, nPR, or PR) until CLL progression or death. DOR analysis will only include responders.
Time to Next Treatment (TTNT) | Up to approximately 70 months
  TTNT is defined as the time from randomization to the start of the next treatment for CLL.
Change from Baseline in Score on European Organization for Research and Treatment of Cancer (EORTC) Item Library (IL)-409 Questionnaire | At baseline and up to approximately 70 months
  Patient-reported symptoms of global health status (GHS), role functioning, and physical functioning, symptom burden and physical condition/fatigue will be measured using the European Organization for Research and Treatment of Cancer quality of life questionnaire EORTC IL-409 (an itemized version of [EORTC] quality of life questionnaire core 30 [QLQ-C30] and its CLL module CLL17). The EORTC-IL-409 consists of 17 questions answered on a 4-point scale where 1 = Not at all (best) to 4 = Very Much (worst) and 2 global health questions answered on a 7-point scale where 1 = Very poor (worst) to 7 = Excellent (best). Higher scores in GHS and functional scales and lower scores in symptom scales indicate better quality of life.

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Study Director — BeOne Medicines

IPD SHARING:
Plan to Share IPD: Yes
BeOne shares data on completed studies responsibly and provides qualified scientific and medical researchers access to data and supporting documentation for clinical trials in dossiers for medicines and indications after submission and approval in the United States, China, and Europe. Clinical trials supporting subsequent local approvals, new indications, or combination products are eligible for sharing once corresponding regulatory approvals are achieved.
  BeOne shares data only when permitted by applicable data privacy and security laws and regulations, when it is feasible to do so without compromising the privacy of study participants, and other considerations.
  Qualified researchers with appropriate competencies who are engaged in novel scientific research may submit a request for participant-level data with a research proposal for BeOne review. Research teams must include a biostatistician and sign a Data Sharing Agreement prior to receiving access to clinical trial data.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: See plan description
Access Criteria: See plan description
URL: https://beonemedicines.com/science/clinical-trials/